CLINICAL TRIAL: NCT06289231
Title: Possibility of Using a Mobile Application for Three-plane Gait Analysis.
Brief Title: The Use of Artificial Intelligence (AI) for Gait Analysis
Status: Not yet recruiting | Type: Observational
Sponsor: Gdansk University of Physical Education and Sport (Other)
Responsible Party: Sponsor
Other Study IDs: AWFiS/2023_5_PE
Record Dates: First submitted 2024-02-19; First posted 2024-03-01 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Gait
Keywords: Vicon; Gait analysis; Artificial intelligence; Tracking movement; Pose estimation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main purpose of this study will be to assess the consistency and reliability of measurements made using the Vicon three-plane gait analysis device (Vicon Motion Capture System Ltd, Oxford, UK) and a mobile application based on image recognition technology with the help of artificial intelligence.

DETAILED DESCRIPTION:
The study will involve 50 healthy, physically active people aged 20-25. The participants will be subjected to movement analysis using the Vicon three-plane gait analysis system using reflective markers. Each of them will make 6 walks at their natural pace along a 10 m long path, during which a three-plane image of their walking will be recorded by the Vicon system. Additionally, during the examination, video recording of the full gait cycle in the sagittal plane from both sides, in the front plane from both sides and at an angle of 30, 45 and 60 degrees will be made using a smartphone camera. The recorded gait cycle using the camera will be analyzed in an image recognition application, which will generate angular values of the lower limb joints. First, the values generated by the Vicon system and the application from the sagittal plane recording will be compared. Then, the consistency of the values generated by the application from the recordings in the sagittal plane on both sides for the same lower limb will be checked. The last step will be to compare the compliance of the angular values from the Vicon system with the data generated in the application from recordings at angles of 60, 45, 30 and 0 degrees.

ELIGIBILITY:
Inclusion Criteria:

* healthy people aged 20-25 years

Exclusion Criteria:

* orthopaedic disease
* neurological disease
* rheumatological disease
* pain in lower limbs in the last 6 months
* pain in lumbar spine in the last 6 months
* surgeries of lower limbs in the last 6 months
* surgeries of spine in the last 6 months
* musculoskeletal injuries in the lower limbs in the last 6 months
* musculoskeletal injuries in the lumbar spine in the last 6 months
* overweight and obesity, determined on the basis of the BMI value

Ages: 20 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Students of the Academy of Physical Education and Sport in Gdańsk,
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Gait analysis by the Vicon system | 45 minutes
  To perform gait analysis, it is necessary to attach reflective markers to the subject at specific anthropometric points. Participants will be asked to walk barefoot in a relaxed manner at a self-selected comfort speed through a 10-meter path (6 repetitions of walking). Each passage through the path will be recorded using the Vicon three-plane gait assessment system, which generates angular values of the ankle, knee and hip joints (degree).
Gait analysis by the mobile image recognition application | 45 minutes
  During the gait analysis using the Vicon system, video recording of the full gait cycle in the sagittal plane from both sides, in the front plane from both sides and at an angle of 30, 45 and 60 degrees will be made using a smartphone camera. The recorded gait cycle using the camera will be analyzed in an image recognition application, which will generate angular values of the lower limb joints (degree).

CONTACTS AND LOCATIONS:
Overall Officials: Paulina W Ewertowska, PhD, Study Chair — Gdansk University of Physical Education and Sport
Locations (1):
- Gdansk University of Physical Education and Sport, Gdansk, Pomeranian Voivodeship, Poland